CLINICAL TRIAL: NCT06479993
Title: The Influence of Chlorella Supplementation on Running Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 21745/002.1
Record Dates: First submitted 2024-02-02; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-02

CONDITIONS: Athletes; Healthy
Keywords: Running; VO2max; Lactate; Oxygen Consumption

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorella supplementation (Experimental): Supplementation of chlorella (6g/day for 3-weeks)
  Interventions: Dietary Supplement: Chlorella supplementation
- Placebo supplementation (Placebo Comparator): Supplementation of placebo (6g/day for 3-weeks)
  Interventions: Dietary Supplement: Placebo supplementation

INTERVENTIONS:
Dietary Supplement: Chlorella supplementation — Supplementation with chlorella (6g/day for 3-weeks)
  Arms: Chlorella supplementation
Dietary Supplement: Placebo supplementation — Supplementation with placebo - microcrystalline cellulose (6g/day for 3-weeks)
  Arms: Placebo supplementation

SUMMARY:
Algae, such as chlorella, are gaining popularity as a nutritious additive to whole food or as a supplement. They contain a variety of beneficial nutrients like vitamins, minerals, healthy fats, and amino acids, which can have positive effects on our health and possibly athletic performance. Chlorella, specifically, is a type of single-celled green algae that you can easily find in health stores worldwide. While there's some evidence suggesting that chlorella supplementation might improve submaximal and maximal performance for cyclists, it's unclear if it has the same impact on runners. To investigate this, the investigators aim to conduct a double-blind randomised placebo controlled study to see if taking chlorella daily for 3-weeks can enhance different aspects of running performance, both during low/moderate and intense exercise, among individuals who regularly engage in running.

DETAILED DESCRIPTION:
After signing the consent form, we will invite you to come to the ISEH laboratory on Tottenham Court Road so we can take some basic baseline readings. This should last up to 60 minutes and will also include a V̇o2max Test (visit 1). After this, you will be randomly allocated either start on chlorella or placebo first. After supplementation (for visit 2 and 3) you will be required to perform a submaximal running test which will entail running at 60% GET (gas exchange threshold), 80% GET, and 75% of the change from peak. This will then be shortly followed by an incremental test to fatigue.

You will then be required to undergo the exact same supplementation period on the alternative supplement with the same exercise test performed.

You will be required to come into the laboratory a total of 3 times. Each visit should take roughly 1 - 1.5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-50.
* Run regularly (3-4 times a week).
* Train with a purpose to compete.
* Consider running to be your main sport.
* Be comfortable running continuously for over 30-minutes at moderate intensity.
* Represent a local running club.

Exclusion Criteria:

* Individuals taking blood thinners.
* Known allergies to algae/mould and iodine.
* Any illness/conditions identified on PARQ (please see attached PARQ)
* Taking immunosuppressant medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Changes in maximal oxygen uptake | Following each 3-week supplementation period of either chlorella or placebo
  Changes in cardiovascular fitness variables as measured by a Cardio Pulmonary Exercise Test following the submaximal run.
Changes in oxygen consumption and oxygen cost | Following each 3-week supplementation period of either chlorella or placebo
  Assessing the possible changes in oxygen consumption and oxygen cost (ml/kg/min) at 60% Gas Exchange threshold (GET), 80% GET, and 75% change as measured by a metabolic cart (Vyntus)
Changes in the respiratory exchange ratio | Following each 3-week supplementation period of either chlorella or placebo
  Assessing the possible changes in the respiratory exchange ratio at 60% Gas Exchange threshold (GET), 80% GET, and 75% change as measured by a metabolic cart (Vyntus)
Changes in heart rate | Following each 3-week supplementation period of either chlorella or placebo
  Assessing the possible changes in heart rate (bpm) at 60% Gas Exchange threshold (GET), 80% GET, and 75% change as measured by a metabolic cart (Vyntus)
Changes in lactate | Following each 3-week supplementation period of either chlorella or placebo
  Assessing the possible changes in blood lactate at 60% Gas Exchange threshold (GET), 80% GET, and 75% change, at maximal oxygen uptake, and 15-mins post maximal as measured by the Biosen.
Changes in glucose | Following each 3-week supplementation period of either chlorella or placebo
  Assessing the possible changes in blood glucose at 60% Gas Exchange threshold (GET), 80% GET, and 75% change, at maximal oxygen uptake, and 15-mins post maximal as measured by the Biosen.

SECONDARY OUTCOMES:
Changes in nutritional status | Following each 3-week supplementation period of either chlorella or placebo
  Assessing the possible changes in nutritional status (macro and micronutrient intake) as measured by food recall.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Gurney, Principal Investigator — University College, London
Locations (1):
- University Colllege London (ISEH), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No